CLINICAL TRIAL: NCT01134588
Title: Assessment of Quality of Life in Disorders of the Pelvic Floor
Acronym: U-GYN-QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LOCAL/2009/VL-01
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference group (Active Comparator): This group will fill out paper questionnaires.
  Interventions: Other: Paper questionnaire
- Experimental group (Experimental): This group will fill out touch-screen questionnaires.
  Interventions: Other: Touch screen questionnaire

INTERVENTIONS:
Other: Paper questionnaire
  Arms: Reference group
Other: Touch screen questionnaire
  Arms: Experimental group

SUMMARY:
The purpose of this study is to compare the touch-screen version of the PFDI-20, PFIQ-7, PISQ 12 and SF-36 french questionnaires to their paper versions. The investigators hypothesize that the percentage of completely filled questionnaires will be higher in the touch-screen version.

ELIGIBILITY:
Inclusion Criteria:

* the patient has pelvic organ prolapse
* the patient requires a surgical intervention within the next 4 to 8 weeks
* the patient understands and reads french
* the patient is affiliated with a social security system
* the patient has given consent

Exclusion Criteria:

* the patient refuses to participate
* the patient is under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Presence / absence of a completely filled out questionnaire | 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, France